CLINICAL TRIAL: NCT01122498
Title: A Phase 1, Randomized, Open-Label, Standard Of Care Control, Dose-Escalating, Multicenter, Safety Study Of BMP-655/ACS As An Adjuvant Therapy For Treatment Of Full-Thickness Rotator Cuff Tears Treated By Means Of An Open Surgical Repair
Brief Title: A Safety Study Of BMP-655/ACS As An Adjuvant Therapy For Treatment Of Rotator Cuff Tears
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3202V1-1003; B1861003
Record Dates: First submitted 2010-05-03; First posted 2010-05-13 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: BMP-655/ACS+Standard of care or Standard of care
- 2 (Experimental)
  Interventions: Biological: BMP-655/ACS+Standard of care or Standard of care
- 3 (Experimental)
  Interventions: Biological: BMP-655/ACS+Standard of care or Standard of care

INTERVENTIONS:
Biological: BMP-655/ACS+Standard of care or Standard of care — BMP-655/ACS 0.015mg/mL
  Arms: 1
Biological: BMP-655/ACS+Standard of care or Standard of care — BMP-655/ACS 0.05mg/mL
  Arms: 2
Biological: BMP-655/ACS+Standard of care or Standard of care — BMP-655/ACS 0.15mg/mL or 0.025mg/mL
  Arms: 3

SUMMARY:
Subjects undergoing an open surgical repair for their torn Rotator Cuff (RC) will be consented, screened, and enrolled in the study if they meet all eligibility criteria. At the time of open surgical repair, subjects who are randomized to receive the test article in addition to the Standard of Care (SOC) will be hospitalized and have a single dose of BMP-655/ACS surgically implanted at the site of tendon attachment to bone. Subjects who are randomized to receive SOC alone will receive no test article. Following surgery, subjects will be prescribed a rehabilitation plan. Subjects will then complete 9 follow-up visits beginning 24 hours after surgery and continuing through 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male subjects and surgically sterile or postmenopausal Japanese female subjects between the ages of 25 and 75 years.
* without tears of the subscapularis or labral pathology requiring surgical repair, as estimated on closed magnetic resonance imaging (MRI) within 3 months before surgery.
* In the shoulder under study, subjects should be able to achieve a passive range of motion (ROM), which is at least 150 degrees in forward elevation (flexion), abduction, and elevation in the scapular plane (scapular abduction). Subjects should have at least 40 degrees of passive ROM in external rotation. In the contralateral shoulder, subjects should be able to achieve active ROM, which is at least 150 degrees in forward elevation (flexion), abduction, and elevation in the scapular plane (scapular abduction). Subjects should have at least 40 degrees of active ROM in external rotation.

Exclusion Criteria:

* Subjects who have had previous surgical intervention to the shoulder joint under study (eg, shoulder arthroscopy, acromioplasty, previous RCR, fracture). Subjects with stage 3 or 4 fatty infiltration (according to the Goutallier grading scale) of their RC muscles on MRI taken within 3 months prior to surgical repair or subjects with moderate or severe degenerative glenohumeral arthritis (according to the Samilson and Prieto arthrosis grading scale ), avascular necrosis, calcific tendonitis, chondrocalcinosis, hypertrophic osteoarthropathy, or Paget disease of the shoulder under study or any bone abnormalities (eg, HO, previous fracture) as confirmed on a radiograph within 3 months prior to surgical repair.
* Subjects with rheumatologic conditions (eg, rheumatoid arthritis, ankylosing spondylitis) affecting the shoulder joints, or autoimmune disorders. Subjects treated with more than 3 corticosteroid injections in the shoulder under study within 1 year prior to planned surgery or subjects treated with any corticosteroid injection in the shoulder under study within 3 months prior to planned surgery or subjects currently receiving oral corticosteroids or taking them within the past 3 months.
* Subjects who are either unwilling or unable (eg, because of claustrophobia or the presence of an automatic cardioverter defibrillator) to undergo examination with closed MRI. Subjects with any other major illness/condition that will substantially increase the risk associated with the subject's participation in and completion of the study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Assess the safety and tolerability of 3 concentrations of BMP-655/ACS in Japanese subjects with full-thickness RCTs treated by means of an open surgical repair. | 12, 26 and 52 weeks

SECONDARY OUTCOMES:
Assess the feasibility of implanting BMP-655/ACS through an open surgical procedure in Japanese subjects and detect circulating levels of BMP-655 in the blood of Japanese subjects. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- Japan (9):
  - Pfizer Investigational Site, Chikushino-shi, Fukuoka
  - Pfizer Investigational Site, Kure, Hiroshima
  - Pfizer Investigational Site, Koushi, Kumamoto
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Toyonaka, Osaka
  - Pfizer Investigational Site, Hiroshima
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Kumamoto
  - Pfizer Investigational Site, Nagano

REFERENCES:
- [Derived] Ide J, Mochizuki Y, van Noort A, Ochi H, Sridharan S, Itoi E, Greiner S. Local rhBMP-12 on an Absorbable Collagen Sponge as an Adjuvant Therapy for Rotator Cuff Repair-A Phase 1, Randomized, Standard of Care Control, Multicenter Study: Part 2-A Pilot Study of Functional Recovery and Structural Outcomes. Orthop J Sports Med. 2017 Sep 12;5(9):2325967117726740. doi: 10.1177/2325967117726740. eCollection 2017 Sep. PMID 28932752